CLINICAL TRIAL: NCT06720740
Title: The RELIEF™ Ureteral Stent - Assessment of Retrograde Urinary Reflux
Brief Title: The RELIEF™ Ureteral Stent Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: The Ureteral Stent Company (Unknown)
Responsible Party: Principal Investigator, Seth Bechis, Associate Professor of Urology, University of California, San Diego
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 809792
Record Dates: First submitted 2024-11-25; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Kidney Stone
Keywords: ureteral stent
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Standard of Care Ureteral Stent (Active Comparator)
  Interventions: Device: Standard of Care Ureteral Stent
- RELIEF Ureteral Stent (Experimental)
  Interventions: Device: RELIEF Ureteral Stent

INTERVENTIONS:
Device: RELIEF Ureteral Stent — The study intervention is placement of the RELIEF Ureteral Stent
  Arms: RELIEF Ureteral Stent
Device: Standard of Care Ureteral Stent — The control product is the Ascerta stent by Boston Scientific.
  Arms: Standard of Care Ureteral Stent

SUMMARY:
Assessment of the backwards flow of urine from the bladder into the ureter (retrograde urine reflux) after placement of the RELIEF® Ureteral Stent using imaging of the bladder after filling it with contrast and assigning a urinary reflux grade. Randomized controlled trial for evaluation of the stent placement and the adequacy of short term drainage (defined as the presence of the stent in the ureter and the lack of surgical or standard of care double J stent to treat symptoms associated with the stent itself on the stented side during the first 48 hours).

ELIGIBILITY:
Inclusion Criteria:

* Has capacity to consent
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Persons, 18 years of age or older
* Male or female subjects with confirmed ureteral and/or renal stones or strictures documented via abdomen X-ray KUB (kidney ureter bladder) or CT (computed tomography)

Exclusion Criteria:

* Distal ureteral obstruction where suture portion of stent may be placed
* Urinary reflux (assessed by pre-stent cystogram)
* Pregnancy or lactation
* Patients requiring bilateral surgical stone management procedure
* Infected stones
* Patients where 24cm or 26cm stent lengths are not suitable
* Ureteral structure in distal third of ureter
* Intraoperative exclusion: based on urologist's discretion, if trauma has been induced to the distal ureter due to ureteroscopy maneuvers, exclude these patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Retrograde urine reflux | At time of stent placement - Day 0, and through study completion - an average of 12 weeks post-operatively
  Assessment of retrograde urine reflux after placement of a ureteral stent using cystography after contrast gravity-filling of the bladder and assigning a urinary reflux grade based on standard scoring.

SECONDARY OUTCOMES:
Stent symptoms | Up until stent removal - Day 7-14, and through study completion - and average of 12 weeks post-operatively
  Assessment of stent symptoms (incidence, relationship to device, severity) attributed to the ureteral stent; Reporting the Ureteral Stent Symptoms Questionnaire (USSQ) before stent placement, after placement at day 3, prior to removal and post removal; Visualization of distal coil floating in bladder (Y/N) after stent placement

CONTACTS AND LOCATIONS:
Overall Officials: Seth K Bechis, MD, Principal Investigator — University of California, San Diego

REFERENCES:
- [Background] Chew BH, Knudsen BE, Denstedt JD. The use of stents in contemporary urology. Curr Opin Urol. 2004 Mar;14(2):111-5. doi: 10.1097/00042307-200403000-00011. PMID 15075840
- [Background] Joshi HB, Okeke A, Newns N, Keeley FX Jr, Timoney AG. Characterization of urinary symptoms in patients with ureteral stents. Urology. 2002 Apr;59(4):511-6. doi: 10.1016/s0090-4295(01)01644-2. PMID 11927301
- [Background] Chambade D, Thibault F, Niang L, Lakmichi MA, Gattegno B, Thibault P, Traxer O. [Study of the safety of double J ureteric stents]. Prog Urol. 2006 Sep;16(4):445-9. French. PMID 17069037
- [Background] Shao Y, Shen ZJ, Zhuo J, Liu HT, Yu SQ, Xia SJ. The influence of ureteral stent on renal pelvic pressure in vivo. Urol Res. 2009 Aug;37(4):221-5. doi: 10.1007/s00240-009-0199-z. Epub 2009 Jun 10. PMID 19513705
- [Background] Giannarini G, Keeley FX Jr, Valent F, Manassero F, Mogorovich A, Autorino R, Selli C. Predictors of morbidity in patients with indwelling ureteric stents: results of a prospective study using the validated Ureteric Stent Symptoms Questionnaire. BJU Int. 2011 Feb;107(4):648-54. doi: 10.1111/j.1464-410X.2010.09482.x. PMID 20590539
- [Background] Krebs A, Deane LA, Borin JF, Edwards RA, Sala LG, Khan F, Abdelshehid C, McDougall EM, Clayman RV. The 'buoy' stent: evaluation of a prototype indwelling ureteric stent in a porcine model. BJU Int. 2009 Jul;104(1):88-92. doi: 10.1111/j.1464-410X.2008.08338.x. Epub 2009 Jan 14. PMID 19154469

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-24): https://cdn.clinicaltrials.gov/large-docs/40/NCT06720740/Prot_SAP_000.pdf
  • Informed Consent Form (2024-07-24): https://cdn.clinicaltrials.gov/large-docs/40/NCT06720740/ICF_001.pdf